CLINICAL TRIAL: NCT00927264
Title: A+ Head Start Intervention for Smoke Free Homes
Brief Title: PRIDE: Preventing Respiratory Illnesses During Childhood Study
Acronym: PRIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: 664; R18HL092901-01 (NIH)
Record Dates: First submitted 2009-06-23; First posted 2009-06-24 (Estimated); Results first posted 2017-08-24 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Tobacco Smoke Pollution
Keywords: tobacco smoke exposure smoking
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Who Masked: Investigator
Masking Description: For masking we were unable to mask the caregiver and child participant since they knew if they were receiving intervention component. The investigator was masked, but outcome assessor may have known group assignment.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral (Experimental): Motivational Interviewing Intervention Plus Education
  Caregivers will receive a home-based motivational interviewing intervention for ETS reduction plus an educational program for ETS reduction.
  Interventions: Behavioral: Motivational Interviewing Intervention for ETS Reduction
- Education Only (Active Comparator): Caregivers will receive only educational program for ETS reduction.
  Interventions: Behavioral: Educational Program for ETS Reduction

INTERVENTIONS:
Behavioral: Motivational Interviewing Intervention for ETS Reduction — The intervention is designed to motivate caregivers to reduce a child's ETS exposure by establishing a complete home and car smoking ban and by considering smoking cessation. Caregivers will receive 2 home visits & 2 telephone session, both with a health counselor. Caregivers will be provided with feedback on air nicotine levels and child salivary cotinine levels. The main target for the intervention will be the primary caregiver of the child because the primary caregiver is ultimately responsible for protecting the child from ETS exposure. Any and all household members may participate in the intervention visits but are not required to do so.
  Arms: Behavioral
Behavioral: Educational Program for ETS Reduction — An Environmental Protection Agency-based educational program that will consist of information about reducing tobacco smoke exposure.
  Arms: Education Only

SUMMARY:
Environmental tobacco smoke (ETS0, also known as secondhand smoke, is the combination of smoke given off by the burning end of a tobacco product and the smoke exhaled by the smoker. Children exposed to ETS are at an increased risk of sudden infant death syndrome (SIDS), ear infections, colds, pneumonia, bronchitis and more severe asthma. ETS can also slow the growth of children's lungs and can cause them to cough, wheeze and fell breathless. The purpose of this study is to determine the effectiveness of a motivational interviewing-based program in reducing ETS exposure and improving lung health among children who are enrolled in a Head Start program and whose households include a smoker.

DETAILED DESCRIPTION:
About 90% of nonsmoking people in the US are exposed to ETS. More than 50 chemicals identified in ETS have been found to cause cancer and exposure has been linked to heart disease in adults and SIDS, ear infections and numerous respiratory problems, including asthma in children. In 2007, the Environmental Protection Agency and the Office of Head Start-a national program that provides economically disadvantaged children services to enhance their social and cognitive development-announced a new initiative to promote smoke-free homes for children in Head Start programs. Because Head Start reaches high-risk, low-income preschool children, it offers a timely intervention for reducing children's exposure to ETS. Head Start also attempts to engage parents, which is an important component of reducing household ETS exposure among children. This study will determine the effectiveness of a home-delivered, motivational interviewing-based program in reducing ETS exposure and improving lung health among children who are enrolled in the Baltimore City Head Start program and whose households include a smoker.

Participation in this study will last 1 year. First, all participating families will be visited at home by a study staff person who will attach special filters that will track the amount of nicotine in the various rooms of the house. During this initial visit, the participating children will undergo weight and height measurements and saliva sampling. About a week later, the filters will be collected, a 2nd saliva samples will be taken and parents will be interviewed about their family and child's health. Families will then be randomly assigned to one of two groups. Both groups will received educational information about reducing tobacco smoke exposure. One group will also receive the home-delivered, motivational interviewing-based program aimed to reduce ETS. This program will consist of 2 home visits and 2 phone calls, both led by health counselor who will teach participants how to reduce their child's exposure to tobacco smoke. The home visits will occur during Weeks 1 & 2 and the phone calls will occur during Weeks 3 & 6. Follow-up visits for all participating families will occur at Months 3,6 and 12 and will involve repeat filter testing, saliva monitoring and interviews.

ELIGIBILITY:
Inclusion Criteria:

* Child enrolled in Baltimore City Head Start
* Smoker living in the home with child

Exclusion Criteria:

* No smoker in home with child
* Does not speak English
* Is enrolled in other respiratory research study

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 350 (Actual)
Dates: Start 2009-01; Primary Completion 2013-01 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia S Rand, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
We will not be sharing individual participant data

REFERENCES:
- [Result] Eakin MN, Rand CS, Borrelli B, Bilderback A, Hovell M, Riekert KA. Effectiveness of motivational interviewing to reduce head start children's secondhand smoke exposure. a randomized clinical trial. Am J Respir Crit Care Med. 2014 Jun 15;189(12):1530-7. doi: 10.1164/rccm.201404-0618OC. PMID 24821270

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Caregivers of children were recruited from 16 Baltimore City Head Start programs from April 2009 to August 2012 with final data collection ending August 2013.
Pre-assignment Details: Caregivers had to complete a baseline assessment prior to randomization and reported information for themselves and the targeted child due to the young age of the child. 350 caregivers were recruited but only 330 were randomized because 20 did not complete the baseline assessment.
Groups:
- Behavioral: Motivational Interviewing Intervention Plus Education
  Participants will receive a home-based motivational interviewing intervention for ETS reduction plus an educational program for ETS reduction.
  Motivational Interviewing Intervention for ETS Reduction: The intervention is designed to motivate families to reduce a child's ETS exposure by establishing a complete home and car smoking ban and by considering smoking cessation. Families will receive 2 home visits & 2 telephone session, both with a health counselor. Families will be provided with feedback on air nicotine levels and child salivary cotinine levels. The main target for the intervention will be the primary caregiver of the child because the primary caregiver is ultimately responsible for protecting the child from ETS exposure. Any and all household members may participate in the intervention visits but are not required to do so.
- Education Only: Participants will receive only educational program for ETS reduction.
  Educational Program for ETS Reduction: An Environmental Protection Agency-based educational program that will consist of information about reducing tobacco smoke exposure.
Period: Overall Study
Arm/Group | Behavioral | Education Only
Started | 165 | 165
Completed | 109 | 140
Not Completed | 56 | 25

BASELINE CHARACTERISTICS:
Population: Eligible caregivers had to be the parent or legal guardian of a child aged 6 months to 6 years, who reported one or more smokers living in the home, and who spoke English. The enrolled caregiver did not have to be the smoker.
Groups:
- Behavioral: Motivational Interviewing Intervention Plus Education
  Caregivers of children will receive a home-based motivational interviewing intervention for ETS reduction plus an educational program for ETS reduction.
  Motivational Interviewing Intervention for ETS Reduction: The intervention is designed to motivate caregivers to reduce a child's ETS exposure by establishing a complete home and car smoking ban and by considering smoking cessation. Caregivers will receive 2 home visits & 2 telephone session, both with a health counselor. Caregivers will be provided with feedback on air nicotine levels and child salivary cotinine levels. The main target for the intervention will be the primary caregiver of the child because the primary caregiver is ultimately responsible for protecting the child from ETS exposure. Any and all household members may participate in the intervention visits but are not required to do so.
- Total: Total of all reporting groups
Arm/Group | Behavioral | Education Only | Total
Number analyzed (Participants) | 165 | 165 | 330
Age, Continuous [Mean (Standard Deviation); unit: years]
  child age | 3.81 (0.81) | 3.71 (.82) | 3.76 (0.82)
  caregiver age | 32.07 (8.6) | 32.12 (9.18) | 32.09 (8.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Child Gender: Female | 87 | 78 | 165
  Child Gender: Male | 78 | 87 | 165
  Caregiver Gender: Female | 140 | 148 | 288
  Caregiver Gender: Male | 25 | 17 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race of child enrolled in study
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 0 | 0
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 153 | 149 | 302
    White | 10 | 9 | 19
    More than one race | 2 | 7 | 9
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Participant unit of measure is child + consented caregiver
  participants
    United States | 165 | 165 | 330

OUTCOME MEASURES:

1. Primary Outcome: Air Nicotine Levels
Description: Air nicotine levels were an indicator of child's exposure to environmental tobacco smoke (ETS)
Time Frame: Measured at Baseline, 3, 6 and 12 months
Population: The number analyzed differs at each time point due to missing data. Reasons for missing data include unable to contact
Measure: Median (Inter-Quartile Range); unit: mg/m^3
Arm/Group | Behavioral | Education Only
Number analyzed (Participants) | 165 | 165
mg/m^3
  Baseline: number analyzed (Participants) | 164 | 164
  Baseline | 1.17 [0.24 to 2.92] | 0.58 [0.08 to 2.01]
  3 month: number analyzed (Participants) | 122 | 134
  3 month | 0.71 [0.22 to 1.88] | 0.51 [0.06 to 1.71]
  6 month: number analyzed (Participants) | 111 | 128
  6 month | 0.75 [0.22 to 2.07] | 0.52 [0.05 to 1.61]
  12 month: number analyzed (Participants) | 105 | 132
  12 month | 0.55 [0.07 to 1.37] | 0.32 [0.04 to 1.5]

2. Secondary Outcome: ETS Reduction, as Measured by Child's Cotinine Levels
Description: Child salivary cotinine will be a measure to evaluate environmental tobacco smoke (ETS) reduction
Time Frame: Measured at Baseline, 3, 6 and 12 months
Population: The number analyzed differs at each time point due to missing data. Reasons for missing include unable to contact, samples not able to be analyzed due to insufficient quantity of saliva collected, or child not available during assessment.
Measure: Median (Inter-Quartile Range); unit: ng/mL
Arm/Group | Behavioral | Education Only
Number analyzed (Participants) | 165 | 165
ng/mL
  Baseline: number analyzed (Participants) | 162 | 162
  Baseline | 4.14 [1.8 to 7.5] | 3.00 [1.34 to 6.26]
  3 Months: number analyzed (Participants) | 123 | 136
  3 Months | 4.14 [1.63 to 6.97] | 3.25 [1.24 to 6.41]
  6 Months: number analyzed (Participants) | 117 | 138
  6 Months | 3.60 [1.55 to 7.40] | 3.04 [1.32 to 5.92]
  12 Months: number analyzed (Participants) | 111 | 139
  12 Months | 4.04 [2.13 to 7.17] | 2.83 [1.37 to 6.07]

3. Secondary Outcome: Respiratory Function of Child by Self Report of Parent
Description: Number of cold infections child experienced in previous 3 months, reported by caregiver
Time Frame: Measured at Baseline, 3, 6, and 12 months
Population: The number analyzed differs at each time point due to missing data. Reasons for missing include unable to contact or caregiver refused or did not fully complete survey
Measure: Mean (Standard Deviation); unit: cold infections
Arm/Group | Behavioral | Education Only
Number analyzed (Participants) | 165 | 165
cold infections
  Baseline: number analyzed (Participants) | 164 | 165
  Baseline | 1.07 (1.06) | 1 (1.00)
  3 Months: number analyzed (Participants) | 126 | 138
  3 Months | 0.44 (0.56) | 0.54 (0.88)
  6 Months: number analyzed (Participants) | 121 | 140
  6 Months | 0.38 (0.65) | 0.36 (0.52)
  12 Months: number analyzed (Participants) | 109 | 140
  12 Months | 0.32 (0.77) | 0.33 (0.51)

4. Secondary Outcome: Health Care Utilization by Child- Self Report From Parent/Caregiver
Description: Parent caregiver reported urgent care visits, number of hospitalizations, and number of emergency department visits in the 12 months prior for child enrolled in study
Time Frame: Measured at baseline and 3, 6 and 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral | Education Only
Number analyzed (Participants) | 165 | 165
Participants
  BL Urgent Care Visits | 80 | 73
  3M Urgent Care Visits | 18 | 15
  6M Urgent Care Visits | 14 | 19
  12M Urgent Care Visits | 13 | 14
  BL Hospitalizations | 10 | 14
  3M Hospitalizations | 4 | 3
  6M Hospitalizations | 1 | 2
  12M Hospitalizations | 1 | 2
  BL Emergency Dept Visit | 75 | 74
  3M Emergency Dept Visit | 18 | 13
  6M Emergency Dept Visit | 13 | 13
  12M Emergency Dept Visit | 9 | 14

5. Secondary Outcome: Number of Participants Who Report Endorsing a Home Smoking Ban
Description: Number of participants endorsing presence of home smoking ban
Time Frame: Measured at baseline, 3, 6 and 12 months
Population: The number analyzed differs at each time point due to missing data. Reasons for missing data include unable to contact
Measure: Count of Participants; unit: Participants
Arm/Group | Behavioral | Education Only
Number analyzed (Participants) | 165 | 165
Participants
  BL: number analyzed (Participants) | 163 | 165
  BL | 129 | 118
  3M: number analyzed (Participants) | 126 | 138
  3M | 80 | 89
  6M: number analyzed (Participants) | 121 | 140
  6M | 78 | 83
  12M: number analyzed (Participants) | 109 | 140
  12M | 65 | 82

ADVERSE EVENTS:
Time Frame: Adverse events were collected for enrolled parent/caregiver and child enrolled in study for the duration of their enrollment (1 year)
Arm/Group | Behavioral | Education Only
Serious Adverse Events (participants affected / at risk) | 1/165 | 1/165
Other Adverse Events (participants affected / at risk) | 13/165 | 10/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral (N=165) | Education Only (N=165)
Asthma Hospitalization (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) — asthma exacerbation
Broken Leg Hospitalization (Surgical and medical procedures) | 0 (0) | 1 (1) — broken leg
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Behavioral (N=165) | Education Only (N=165)
Family Stress Related to Smoking (Social circumstances) | 13 (13) | 10 (10) — Parent/caregiver may discuss smoking exposure with others in household- we expect that this may have caused some sources of stress

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No